CLINICAL TRIAL: NCT04556617
Title: A Multicenter, Open-Label, Parallel, Phase 1b/2a Study of PLX2853 in Combination With Abiraterone Acetate and Prednisone and Phase 1b/2a Study of PLX2853 in Combination With Olaparib in Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: PLX2853 in Combination With Abiraterone Acetate and Prednisone and in Combination With Olaparib in Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study terminated due to business realignment
Sponsor: Opna Bio LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLX124-04
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: PLX2853; Metastatic Castration-resistant Prostate Cancer; Olaparib; Abiraterone Acetate; Adenocarcinoma; Prostate Cancer
MeSH Terms: conditions — Adenocarcinoma; Prostatic Neoplasms | interventions — olaparib; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1b PLX2853 (20 mg) + Olaparib (Experimental): Phase 1b dose escalation
  Interventions: Drug: PLX2853 20 mg; Drug: Olaparib
- Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone (Experimental): Phase 1b dose escalation
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: PLX2853 40 mg
- Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone (Experimental): Phase 1b dose escalation
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: PLX2853 80 mg
- Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone (Experimental): Phase 2a dose expansion
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: PLX2853 80 mg
- Phase 1b PLX2853 (40 mg) + Olaparib (Experimental): Phase 1b dose escalation
  Interventions: Drug: Olaparib; Drug: PLX2853 40 mg

INTERVENTIONS:
Drug: PLX2853 20 mg — PLX2853 tablets
  Arms: Phase 1b PLX2853 (20 mg) + Olaparib
Drug: Olaparib — Olaparib tablets
  Arms: Phase 1b PLX2853 (20 mg) + Olaparib; Phase 1b PLX2853 (40 mg) + Olaparib
Drug: Abiraterone acetate — Abiraterone acetate tablets
  Arms: Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone; Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone; Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone
Drug: Prednisone — Prednisone (or equivalent) tablets
  Arms: Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone; Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone; Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone
Drug: PLX2853 40 mg — PLX2853 tablets
  Arms: Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone; Phase 1b PLX2853 (40 mg) + Olaparib
Drug: PLX2853 80 mg — PLX2853 tablets
  Arms: Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone; Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone

SUMMARY:
The purpose of this research study is to evaluate safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of the investigational drug PLX2853 in subjects with Metastatic Castration-Resistant Prostate Cancer (mCRPC)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing informed consent.
2. Histologically confirmed adenocarcinoma of the prostate with tumor tissue available for molecular analyses.
3. Eastern Cooperative Oncology Group Performance Status 0 to 1.
4. Adequate organ function as demonstrated following laboratory values.
5. Fertile male subjects with female sexual partners must agree to use a highly effective method of birth control during the study and for 90 days after the last dose of study drug.
6. Except as specified above for organ function, all drug-related toxicity from previous cancer therapy (including ongoing Abiraterone Acetate + Prednisone therapy if applicable) must be resolved (to Grade ≤1 or baseline per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0) prior to study treatment administration (Grade 2: alopecia, hot flashes, decreased libido, or neuropathy is allowed).
7. Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.

Exclusion Criteria:

1. Prior exposure to a bromodomain inhibitor.
2. History of autoimmune hemolytic anemia or autoimmune thrombocytopenia.
3. Clinically significant cardiac disease.
4. Inability to take oral medication or significant nausea and vomiting, malabsorption, or significant small bowel resection that, in the opinion of the Investigator, would preclude adequate absorption.
5. Active known second malignancy with the exception of any of the following:

   * Adequately treated basal cell carcinoma or squamous cell carcinoma of the skin.
   * Adequately treated Stage I cancer from which the subject is currently in remission and has been in remission for ≥2 years.
   * Any other cancer from which the subject has been disease-free for ≥3 years.
6. Subject is participating in any other therapeutic clinical study (observational or registry studies are allowed).
7. Presence of any other medical, psychological, familial, sociological, or geographic condition potentially hampering compliance with the study protocol or would interfere with the study endpoints or the subject's ability to participate in the study in the judgment of the Investigator.
8. Receipt of any anti-cancer therapy prior to Cycle 1 Day 1 with less than protocol defined wash-out with the exception of Abiraterone Acetate (for subjects enrolling into Abiraterone Acetate Combination) and GnRH therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - Karmanos Cancer Institute, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Tennessee Oncology/ Sarah Cannon, Nashville, Tennessee
  - Virginia Cancer Specialist, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Sarah Cannon Research Institute, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b PLX2853 (20 mg) + Olaparib: Dose escalation
  Once daily dosing PLX2853 20 mg
  Twice daily dosing olap 300 mg
- Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone: Dose escalation Once daily dosing of PLX2853 40 mg AA 1000 mg pred 10 mg
- Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone: Dose escalation Once daily dosing of PLX2853 80 mg AA 1000 mg pred 10 mg
- Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone: Dose expansion Once daily dosing PLX2853 80 mg AA 1000 mg pred 10 mg
- Phase 1b PLX2853 (40 mg) + Olaparib: Dose escalation Once daily dosing PLX2853 40 mg
  Twice daily dosing olap 300 mg
Period: Overall Study
Arm/Group | Phase 1b PLX2853 (20 mg) + Olaparib | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (40 mg) + Olaparib
Started | 1 | 5 | 7 | 5 | 1
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 5 | 7 | 5 | 1
Not completed — progressive disease | 0 | 2 | 2 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 1 | 0
Not completed — PSA increase | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor study termination | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1b PLX2853 (20 mg) + Olaparib: Once daily dosing PLX2853 20 mg
  Twice daily dosing olap 300 mg
- Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone: Once daily dosing of PLX2853 40 mg AA 1000 mg pred 10 mg
- Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone; Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone: Once daily dosing of PLX2853 80 mg AA 1000 mg pred 10 mg
- Phase 1b PLX2853 (40 mg) + Olaparib: Once daily dosing PLX2853 40 mg
  Twice daily dosing olap 300 mg
- Total: Total of all reporting groups
Arm/Group | Phase 1b PLX2853 (20 mg) + Olaparib | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (40 mg) + Olaparib | Total
Number analyzed (Participants) | 1 | 5 | 7 | 5 | 1 | 19
Age, Continuous [Mean (Full Range); unit: years] | 69 [69 to 69] | 66.4 [60 to 78] | 68.9 [58 to 80] | 68.2 [63 to 76] | 73 [73 to 73] | 68.3 [58 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 5 | 7 | 5 | 1 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 2
  White | 1 | 3 | 2 | 3 | 0 | 9
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 1 | 5 | 7 | 5 | 1 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities
Description: Dose limiting toxicity defined as clinically significant adverse events or laboratory abnormalities occurring during first cycle of study drug administration that are possibly related to study drug and that meet specific criteria defined in the protocol
Time Frame: From time of first dose of PLX2853 and combination agent(s) through completion of Cycle 1 (21 days)
Measure: Number; unit: participants
Arm/Group | Phase 1b PLX2853 (20 mg) + Olaparib | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (40 mg) + Olaparib
Number analyzed (Participants) | 1 | 5 | 7 | 5 | 1
participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1b (Both Arms): Incidence of TEAEs That Are Related to Treatment
Description: Treatment-emergent adverse events are those reported after study drug has been administered.
Time Frame: From time of first dose of PLX2853 and combination agent(s) until 30 days from end of treatment (an average of 103 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b PLX2853 (20 mg) + Olaparib | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (40 mg) + Olaparib
Number analyzed (Participants) | 1 | 5 | 7 | 5 | 1
Participants | 1 | 5 | 7 | 5 | 1

3. Primary Outcome: Determination of Maximum Tolerated Dose
Description: To be evaluated in both PLX2853 + AA + pred and PLX2853 + olap group; If DLTs observed in 2 or more subjects the dose will be considered intolerable and MTD will have been reached.
Time Frame: From time of first dose of PLX2853 and combination agent(s) through completion of Cycle 1 (21 days)
Measure: Number; unit: mg
Arm/Group | Phase 1b PLX2853 (20 mg) + Olaparib | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (40 mg) + Olaparib
Number analyzed (Participants) | 1 | 5 | 7 | 5 | 1
mg | NA — Study terminated and MTD not determined as DLTs not observed in 2 subjects or more per protocol definition | NA — Study terminated and MTD not determined as DLTs not observed in 2 subjects or more per protocol definition | NA — Study terminated and MTD not determined as DLTs not observed in 2 subjects or more per protocol definition | NA — Study terminated and MTD not determined as DLTs not observed in 2 subjects or more per protocol definition | NA — Study terminated and MTD not determined as DLTs not observed in 2 subjects or more per protocol definition

ADVERSE EVENTS:
Time Frame: Through 30 days after last study drug, an average of 6 months
Arm/Group | Phase 1b PLX2853 (20 mg) + Olaparib | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone | Phase 1b PLX2853 (40 mg) + Olaparib
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/5 | 0/7 | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/5 | 3/7 | 2/5 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 5/5 | 7/7 | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b PLX2853 (20 mg) + Olaparib (N=1) | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone (N=5) | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone (N=7) | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone (N=5) | Phase 1b PLX2853 (40 mg) + Olaparib (N=1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increase (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b PLX2853 (20 mg) + Olaparib (N=1) | Phase 1b PLX2853 (40 mg) + Abiraterone Acetate + Prednisone (N=5) | Phase 1b PLX2853 (80 mg) + Abiraterone Acetate + Prednisone (N=7) | Phase 2a PLX2853 (80 mg) + Abiraterone Acetate + Prednisone (N=5) | Phase 1b PLX2853 (40 mg) + Olaparib (N=1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (4) | 4 (4) | 7 (7) | 0 (0) | 1 (1)
urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
dry heaving (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 0 (0) | 3 (3) | 6 (6) | 5 (7) | 1 (1)
unsteady gait (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
elevated d-dimer (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
weight loss (Investigations) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
tremors (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
intermittent hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
low appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
itchy skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
worsening hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04556617/Prot_SAP_001.pdf